CLINICAL TRIAL: NCT05840068
Title: Metformin Effect as a Chemotherapeutic Adjuvant on Level of IGF in Non-diabetic Breast Cancer Patients
Brief Title: IGF Level in Breast Cancer Patients Treated With Metformin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Marian S. Boshra, Dr., Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IGF level in breast cancer
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer Female
Keywords: Metformin; Breast cancer; IGF
MeSH Terms: conditions — Breast Neoplasms | interventions — Metformin; Tablets; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin and Chemotherapy (Experimental): Metformin (500 mg twice daily) plus chemotherapy is administered to Group A (n=57)
  Interventions: Drug: MetFORMIN 500 Mg Oral Tablet; Drug: Chemotherapy
- Chemotherapy alone (Other): Chemotherapy is administered alone to Group B (n=50).
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: MetFORMIN 500 Mg Oral Tablet — MetFORMIN 500 Mg Oral Tablet
  Other Names: Glucophage 500 oral tablet and Chemotherapy
  Arms: Metformin and Chemotherapy
Drug: Chemotherapy — The standard chemotherapy protocol developed by the South Egypt Cancer Institute (SECI).
  Other Names: Chemotherapy alone

SUMMARY:
The purpose of this study is to examine the impact of metformin as an adjuvant to chemotherapy on IGF levels in both progressing and non progressing cases of metastatic breast cancer in female patients.

DETAILED DESCRIPTION:
One hundred and seven women with metastatic breast cancer (MBC) are randomly assigned to either a metformin (500 mg twice daily) or placebo (placebo) group during chemotherapy. All patients followed the standard chemotherapy protocol developed by the South Egypt Cancer Institute (SECI). Blood IGF-1 levels were measured at the start of treatment (baseline) and again six months later.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with MBC
* patients older than 18
* nondiabetic patients
* patients who received only chemotherapy

Exclusion Criteria:

* patients with non-metastatic breast cancer
* patients receiving hormonal therapy or radiotherapy
* patients with diabetes
* history of cardiac diseases
* hypersensitivity, or allergy to metformin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 107 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
IGF-1 levels | 6 months.
  IGF-1 levels were measured before and after treatment.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 1 Year
  The measurement values of IGF were divided into two groups, high and low, based on the cut off value. After a year of observation, researchers in both groups compared their progression-free survival (PFS).

CONTACTS AND LOCATIONS:
Locations (1):
- Marian S. Boshra, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ko KP, Ma SH, Yang JJ, Hwang Y, Ahn C, Cho YM, Noh DY, Park BJ, Han W, Park SK. Metformin intervention in obese non-diabetic patients with breast cancer: phase II randomized, double-blind, placebo-controlled trial. Breast Cancer Res Treat. 2015 Sep;153(2):361-70. doi: 10.1007/s10549-015-3519-8. Epub 2015 Aug 21. PMID 26293146
- [Background] Essa NM, Salem HF, Elgendy MO, Gabr A, Omran MM, Hassan NA, Tashkandi HM, Harakeh S, Boshra MS. Efficacy of Metformin as Adjuvant Therapy in Metastatic Breast Cancer Treatment. J Clin Med. 2022 Sep 20;11(19):5505. doi: 10.3390/jcm11195505. PMID 36233373
- [Result] Pollak M. Insulin and insulin-like growth factor signalling in neoplasia. Nat Rev Cancer. 2008 Dec;8(12):915-28. doi: 10.1038/nrc2536. PMID 19029956